CLINICAL TRIAL: NCT01305785
Title: National Registry of Acute Myocardial Infarction in Switzerland
Brief Title: AMIS Plus - National Registry of Acute Myocardial Infarction in Switzerland
Acronym: AMIS Plus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: University of Zurich (Other); University Hospital, Geneva (Other); Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Basel, Switzerland (Other); Triemli Hospital (Other); Kantonsspital Baden (Other); Cantonal Hospital of St. Gallen (Other); University Hospital Freiburg (Other); Cantonal Hospital, Frauenfeld (Other); Hospital Centre Biel/Bienne (Other); Spital Lachen AG (Other); Cardiocentro Ticino (Other)
Responsible Party: Principal Investigator, Prof. Paul Erne, AMIS Plus Steering Committee President, Luzerner Kantonsspital
Other Study IDs: AMIS Plus
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The AMIS Plus national registry collects and analyzes data on patients with acute myocardial infarction in Switzerland in the pre-admission, hospital and follow-up phases. Emphasis is placed on the evaluation of risk factors, diagnostics, urgent therapy strategies and treatment of acute coronary syndrome. The AMIS Plus data gathered are important for assessing guidelines, improving compliance with guidelines in clinical practice, investigating patient groups not extensively studied in large randomized trials, quality assurance as well as the continuous improvement of therapeutic strategies based on a large database.

DETAILED DESCRIPTION:
The AMIS Plus project has two main goals:

1. To Maintain a Nationwide Registry

   * An ongoing nationwide registry (databank) of acute coronary syndromes
   * Description of the patient population with acute coronary syndromes
   * Description of characteristics of treatment and hospitalization
   * Description of outcomes 3- and 12-months after admission for ACS
   * Epidemiological studies, e.g. definition of risk factors of patients with acute coronary syndromes, hospital mortality, time and cost-effective strategies as well as outcome measures
2. Quality Control

   * Evaluation of compliance with guidelines for the medical care of acute coronary syndromes
   * Internal quality control through regular feedback and benchmarking

Methods

All Swiss hospitals admitting patients with acute coronary syndrome are eligible. Data are collected on demographics, risk factors, symptoms, laboratory results, invasive therapy, complications and medication.

Since the start in January 1997, the method of data collection has continuously improved in order to suit the different needs and technological advancements of the participating hospitals. Participants can either complete paper questionnaires and send them directly to the AMIS Plus Data Center at the Institute of Social and Preventive Medicine in Zurich where these questionnaires are then checked and entered online or they can enter data directly online (AMIS online questionnaire). Data security has a high priority. Participant identification (code for hospital and physician) and a password are required to access the data entry form and send data.

ELIGIBILITY:
Inclusion Criteria: Patients who had symptoms within the last 48 hours at hospital admission with a discharge clinical diagnosis of acute myocardial infarction or patients who suffered an acute myocardial infarction in hospital during a hospitalization for other reasons.

Exclusion Criteria: Since January 2012, patients with unstable angina are no longer included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute myocardial infarction definition:
  1. Characteristic ischemic symptoms
  2. ECG changes indicating new ischemia (ST-T changes or new left bundle branch block) or developing pathological Q-waves
  3. A dynamic increase or decrease in biomarker or troponin (I or T) levels above the individual hospital cut-off for MI. The internationally accepted guidelines for troponin levels are set at least one value above the 99th percentile of the upper reference limit (URL). Cut-off levels for either total creatine kinase (CK) or creatine kinase MB fraction (CK-MB) at least twice the upper limit of normal.
Sampling Method: Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 1997-01

CONTACTS AND LOCATIONS:
Overall Officials: Paul Erne, MD, Study Director — AMIS Plus Data Center
Locations (1):
- University of Zurich, Zurich, Switzerland

REFERENCES:
- [Result] Radovanovic D, Erne P. AMIS Plus: Swiss registry of acute coronary syndrome. Heart. 2010 Jun;96(12):917-21. doi: 10.1136/hrt.2009.192302. PMID 20538666
- [Derived] Roberto M, Hoepli A, Cattaneo M, Radovanovic D, Rickli H, Erne P, Pedrazzini GB, Moccetti M. Patients With AMI and Severely Reduced LVEF, a Well-Defined, Still Extremely Vulnerable Population (Insights from AMIS Plus Registry). Am J Cardiol. 2023 Aug 1;200:190-201. doi: 10.1016/j.amjcard.2023.05.027. Epub 2023 Jun 20. PMID 37348272
- [Derived] Roberto M, Radovanovic D, Butta C, Tersalvi G, Krull J, Erne P, Rickli H, Pedrazzini GB, Moccetti M. Dual antiplatelet therapy is under-prescribed in patients with surgically treated acute myocardial infarction. Interact Cardiovasc Thorac Surg. 2021 Oct 29;33(5):687-694. doi: 10.1093/icvts/ivab159. PMID 34171919
- [Derived] Bruggmann C, Iglesias JF, Gex-Fabry M, Fesselet R, Vogt P, Sadeghipour F, Voirol P. Long-Term Quality of Prescription for ST-Segment Elevation Myocardial Infarction (STEMI) Patients: A Real World 1-Year Follow-Up Study. Am J Cardiovasc Drugs. 2020 Feb;20(1):105-115. doi: 10.1007/s40256-019-00361-5. PMID 31300969
- [Derived] Radovanovic D, Seifert B, Roffi M, Urban P, Rickli H, Pedrazzini G, Erne P. Gender differences in the decrease of in-hospital mortality in patients with acute myocardial infarction during the last 20 years in Switzerland. Open Heart. 2017 Nov 14;4(2):e000689. doi: 10.1136/openhrt-2017-000689. eCollection 2017. PMID 29177059
- [Derived] Bertel N, Witassek F, Puhan M, Erne P, Rickli H, Naegeli B, Pedrazzini G, Stauffer JC, Radovanovic D. Management and outcome of patients with acute myocardial infarction presenting with pacemaker rhythm. Int J Cardiol. 2017 Mar 1;230:604-609. doi: 10.1016/j.ijcard.2016.12.047. Epub 2016 Dec 20. PMID 28040280
- [Derived] Schoenenberger AW, Radovanovic D, Windecker S, Iglesias JF, Pedrazzini G, Stuck AE, Erne P; AMIS Plus Investigators. Temporal trends in the treatment and outcomes of elderly patients with acute coronary syndrome. Eur Heart J. 2016 Apr 21;37(16):1304-11. doi: 10.1093/eurheartj/ehv698. Epub 2016 Jan 12. PMID 26757786
- [Derived] Erne P, Radovanovic D, Seifert B, Bertel O, Urban P; AMIS Plus Investigators. Outcome of patients admitted with acute coronary syndrome on palliative treatment: insights from the nationwide AMIS Plus Registry 1997-2014. BMJ Open. 2015 Mar 2;5(3):e006218. doi: 10.1136/bmjopen-2014-006218. PMID 25732032
- [Derived] Wildi K, Cuculi F, Twerenbold R, Marxer T, Rubini Gimenez M, Reichlin T, Haaf P, Monsch R, Marsch S, Hunziker P, Bingisser R, Osswald S, Erne P, Mueller C. Incidence and timing of serious arrhythmias after early revascularization in non ST-elevation myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2015 Aug;4(4):359-64. doi: 10.1177/2048872614557230. Epub 2014 Oct 27. PMID 25348273
- [Derived] Radovanovic D, Seifert B, Urban P, Eberli FR, Rickli H, Bertel O, Puhan MA, Erne P; AMIS Plus Investigators. Validity of Charlson Comorbidity Index in patients hospitalised with acute coronary syndrome. Insights from the nationwide AMIS Plus registry 2002-2012. Heart. 2014 Feb;100(4):288-94. doi: 10.1136/heartjnl-2013-304588. Epub 2013 Nov 1. PMID 24186563
- See also: AMIS Plus Registry — http://www.amis-plus.ch